CLINICAL TRIAL: NCT02886429
Title: Safety and Efficacy of Ultrasound Guided Paravertebral Dexmedetomidine for Postoperative Pain Relief in Video Assisted Thoracoscopy Surgery
Brief Title: Post- Thoracotomy Paravertebral Block
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sayed Kaoud Abd-Elshafy, Associate profossor of anesthesia, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIRB0000871250
Record Dates: First submitted 2016-08-27; First posted 2016-09-01 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Pain, Postoperative
Keywords: dexmedetomidine; bupivacaine; Ultrasound guided paravertebral block; pain; post-thoracotomy
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Bupivacaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Active Comparator): Ultrasound guided paravertebral block with bupivacaine group Thirty patients will be given isobaric bupivacaine 0.5% (0.3ml/kg) via paravertebral route.
  Interventions: Drug: Bupivacaine
- Group B (Active Comparator): Ultrasound guided paravertebral block with bupivacaine and dexmedetomidine group Thirty patients will be given isobaric bupivacaine 0.5% (0.3ml/kg) and dexmedetomidine (1 mcg/kg) via paravertebral route (Bupivacaine plus Dexmedetomidine)
  Interventions: Drug: Bupivacaine; Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Bupivacaine — Ultrasound guided paravertebral block with bupivacaine
  Other Names: Marcaine
Drug: Dexmedetomidine — Ultrasound guided paravertebral block with dexmedetomidine
  Other Names: Precedex
  Arms: Group B

SUMMARY:
Postoperative pain is the most undesired consequence of surgery, and if not managed adequately, can lead to delayed recovery and increased hospital stay. Surveys continue to reveal that postoperative pain is insufficiently managed throughout the first world, let alone in the Third World. An American survey over 20 years showed that only one in four patients had adequate relief of postoperative pain. This has led recovery room protocols to include pain as a fifth vital sign that needs to be addressed before patients are discharged to the ward

DETAILED DESCRIPTION:
This prospective, randomized, double-blinded, parallel assignment clinical trial will be done after receiving approval from the local ethics committee of the Faculty of Medicine, Assiut University. A written informed consent will be taken after discussing a detailed description of the study with the patients.

Patients will be allocated randomly into two equal groups by computer programs and will be contained in sealed opaque envelopes.

Patients will be premedicated with midazolam (0.1mg/kg), 30 min before the operation. Patients will be monitored with ECG, non-invasive blood pressure, heart rate, temperature, oxygen saturation, exhaled CO2 (end tidal capnography), and train of four. In both groups, general anesthesia will be induced with propofol (2mg/kg) and fentanyl (1 mcg/kg). Tracheal intubation will be facilitated with cisatracurium 0.1 mg/kg. Anesthesia will be maintained with isoflurane (1-2 %) and cisatracurium (0.05 mg/kg per dose). Fentanyl (0.5mcg/kg) will be repeated if heart rate (HR) and/or mean arterial pressure (MAP) rise 20 % above baseline values. After the end of anesthesia induction and before surgical procedure Technique of ultrasound guided paravertebral block will be done in both groups.

ELIGIBILITY:
Inclusion Criteria:

1. ASA I, II and III.
2. In the age ranged between 18 up to 60 years.
3. Elective video-assisted thoracoscopy

Exclusion Criteria:

1. ASA IV and V
2. Liver impairment
3. Renal impairment
4. allergy to the drugs used
5. Known contraindication for regional techniques such as:

   * Infection near the site of the needle insertion
   * Coagulopathy
   * Anti-coagulation therapy,

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
post-thoracotomy pain | within first 24 hours after Video Assisted Thoracoscopy Surgery
  5. Pain scores at rest and on coughing will be recorded using visual analogue scale (VAS) pain intensities at rest and during coughing/movement assessed by VAS score. The quality of effective analgesia will be expressed as VAS values derived from the VAS pain score, at rest and during coughing during each assessment period (2 h, at 4, 8 and 24 h).

SECONDARY OUTCOMES:
pulmonary function tests | within first 24 hours after Video Assisted Thoracoscopy Surgery
  done preoperatively and at postoperative period
rescue analgesia | within first 24 hours after Video Assisted Thoracoscopy Surgery
  Consumption of IV rescue analgesia attained with ketorolac tromethamine (30 mg per dose).
sedation score | within first 24 hours after Video Assisted Thoracoscopy Surgery
  Richmond Agitation Sedation Score
nausea, vomiting | within first 24 hours after Video Assisted Thoracoscopy Surgery
  nausea, vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Sayed K Abd-Elshafy, MD, Principal Investigator — Associate professor of anesthesia
Locations (1):
- Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided